CLINICAL TRIAL: NCT04123301
Title: Theta-Burst Stimulation (TBS) in Major Depressive Episodes With Mixed Characteristics in Bipolar and Major Depressive Disorder: a Randomized, Controlled, Double-blind, Parallel-group Clinical Trial of Efficacy, Safety, and Tolerability.
Brief Title: Theta-Burst Stimulation in Major Depressive Episodes With Mixed Characteristics.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ricardo Alberto Moreno, M.D., Ph.D., Principal investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MORENO-2019
Record Dates: First submitted 2019-10-02; First posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Depressive Episode; Depressive Disorder; Bipolar Disorder
Keywords: mixed depression; depressive disorder; bipolar disorder; transcranial magnetic stimulation
MeSH Terms: conditions — Depressive Disorder; Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, parallel-group, 6-week, sham-controlled clinical trial.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Allocation masking will be done through sequentially numbered cards that will determine which group each patient will belong to. The card determines whether the coil to be used will produce actual or simulated stimulation. A secretary who does not participate directly in the research will be responsible for handling the numbered cards to the patient prior to each session. Participants and staff will not fully know the status of allocation groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active TBS Arm (Active Comparator): Patients randomized to this arm will receive active TBS 5 consecutive days of the week (Monday to Friday) in the first 3 weeks and then 2 alternate days of the week (with interval of at least 1 day between sessions) for another 3 weeks.
  Interventions: Device: Active Theta Burst Stimulation (TBS)
- Sham TBS Arm (Sham Comparator): Patients randomized to this arm will receive sham TBS 5 consecutive days of the week (Monday to Friday) in the first 3 weeks and then 2 alternate days of the week (with interval of at least 1 day between sessions) for another 3 weeks.
  Interventions: Device: Sham Theta Burst Stimulation (TBS)

INTERVENTIONS:
Device: Active Theta Burst Stimulation (TBS) — Each session will be comprised of ACTIVE TBS: first, continuous inhibitory stimulation (cTBS) in the right dorsolateral prefrontal cortex followed by intermittent excitatory stimulation (iTBS) in the left dorsolateral prefrontal cortex.
  Arms: Active TBS Arm
Device: Sham Theta Burst Stimulation (TBS) — The sham-TBS sessions will be performed using an identical coil that produces SHAM Stimulation: first, sham continuous inhibitory stimulation (cTBS) in the right dorsolateral prefrontal cortex followed by sham intermittent excitatory stimulation (iTBS) in the left dorsolateral prefrontal cortex.
  Arms: Sham TBS Arm

SUMMARY:
The investigators will perform a double-blind, randomized, sham-controlled clinical trial of theta-burst stimulation (TBS) in mixed depressive episodes of both bipolar and major depressive disorders. Will be selected 90 patients aged 18-65 years with diagnosis of TB (I or II) or MDD in moderate or severe major depressive episode with mixed features. The primary endpoint of efficacy will be a continuous outcome of change in Montgomery-Asberg Depression Rating Scale (MADRS) from baseline to week 3.

DETAILED DESCRIPTION:
INTRODUCTION: Mixed-specifier mood disorders are probably a different subgroup in terms of response to treatment, socio-demographic parameters, course and family history. The investigators will perform a clinical trial of theta-burst stimulation (TBS) in mixed depressive episodes of both bipolar (I and II) and major depressive disorders. METHODS: The study is designed as a randomized, sham-controlled, double-blinded clinical trial evaluating TBS for the treatment of moderate or severe major depressive episodes with mixed features of patients receiving at least one first or second line pharmacological treatment for depressive episodes without adequate response. Ninety adult (18 to 65 yo) patients will be enrolled and submitted to 6-week (comprising 5 consecutive days a week sessions for the first 3 weeks and then 2 days a week for a further 3 week) of inhibitory followed by excitatory TBS in dorsolateral prefrontal cortex. Participants will be assessed using clinical and neuropsychological tests before and after the intervention. The primary outcome is change in Montgomery-Asberg Depression Scale (MADRS) score over time and across groups. Cognitive parameters will also be assessed with neuropsychological tests.

ELIGIBILITY:
Inclusion Criteria:

* Current mixed depression in any mood disorder (bipolar I, bipolar II or major depressive disorder) assessed with Montgomery-Asberg Depression Rating Scale (MADRS) score ≥ 20 points AND Young Mania Rating Scale (YMRS) score ≥ 1 point in 3 or more items.
* Any appropriate first or second line pharmacological regimen in accordance with CANMAT guidelines to treat a major depressive episode in major depressive disorder (Agomelatina 25-50 mg/dia; Bupropiona 150-300 mg/dia; Citalopram 20-40 mg/dia; Desvenlafaxina 50 - 100 mg/dia; Duloxetina 60 - 120mg/dia; Escitalopram 10 - 20 mg/dia; Fluoxetina 20 - 60 mg/dia; Fluvoxamina 100 - 300 mg/dia; Mirtazapina 15 - 45 mg/dia; Paroxetina 20 - 60 mg/dia; Sertralina 50 - 200 mg/dia; Venlafaxina 75 - 225 mg/dia; Vortioxetina 10 - 20 mg/dia; Amitriptilina 150 - 300 mg/dia; Imipramina 150 - 300 mg/dia; Clomipramina 150 - 200 mg/dia; Nortriptilina 75 - 150 mg/dia; Trazodona 150 - 300 mg/dia; Quetiapina 150 - 300mg/dia), bipolar I (Quetiapina 300 - 600 mg/dia; Lítio litemia 0,6 - 1,2 mEq/L; Lamotrigina 100 - 200 mg/dia; Lurasidona 40 - 80 mg/dia; Lítio/Divalproato + Lurasidona; Lítio/Divalproato + Lamotrigina; Olanzapina 5 - 20 mg/dia + Fluoxetina 20 - 60 mg/dia; Divalproato de sódio; Lítio/Divalproato + ISRS/Bupropiona) or bipolar II disorder (Quetiapina 300 - 600 mg/dia; Lítio; Lamotrigina; Bupropiona; Sertralina; Venlafaxina).

Exclusion Criteria:

* Concomitant diagnosis of other neuropsychiatric disorders such as: schizophrenia, dementias, mental retardation, organic mental disorder, or epilepsy;
* Acute suicide ideation (assessed by interview and clinical evaluation);
* Suspected or confirmed pregnancy;
* Women in breastfeeding;
* Severe or unstable clinical disease;
* Specific contraindications to TBS: previous epileptic seizures; change in electroencephalogram at some point in life; previous stroke; previous severe TBI (with neurosurgery); metallic object on head (except mouth) as projectile piece, surgical clip, welding fragments; any implanted device (cardiac pacemaker, intravenous catheter).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-03-08 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale (MADRS) at week 3. | From baseline until week 3.
  Change in Montgomery-Asberg Depression Rating Scale (MADRS) in each patient in both interventional groups. The outcome will be assessed by a continuous change using a mixed models statistic. The scale range is: 0 to 6 - normal/symptom absent; 7 to 19 - mild depression; 20 to 34 - moderate depression; 35 - 60 - severe depression. Reduction is a better and increase is a worse outcome.

SECONDARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale (MADRS) at week 6. | From baseline until week 6.
  Change in Montgomery-Asberg Depression Rating Scale (MADRS) in each patient in both interventional groups. The outcome will be assessed by a continuous change using a mixed models statistic. The scale range is: 0 to 6 - normal/symptom absent; 7 to 19 - mild depression; 20 to 34 - moderate depression; 35 - 60 - severe depression. Reduction is a better and increase is a worse outcome.
Change in Young Mania Rating Scale (YMRS) at week 3. | From baseline until week 3.
  Change in Young Mania Rating Scale (YMRS) in each patient in both interventional groups. The outcome will be assessed by a continuous change using a mixed models statistic. The scale range is: 13-19 - hypomania; 20-25 - mild mania; 26-37 - moderate mania ; 38-60 - severe mania. Reduction is a better and increase is a worse outcome.
Change in Young Mania Rating Scale (YMRS) at week 6. | From baseline until week 6.
  Change in Young Mania Rating Scale (YMRS) in each patient in both interventional groups. The outcome will be assessed by a continuous change using a mixed models statistic. The scale range is: 13-19 - hypomania; 20-25 - mild mania; 26-37 - moderate mania ; 38-60 - severe mania. Reduction is a better and increase is a worse outcome.
Response rate using Montgomery-Asberg Depression Rating Scale (MADRS) at week 3 | From baseline until week 3.
  Reduction of 50% or more of the Montgomery-Asberg Depression Rating Scale (MADRS) in each patient in both interventional groups. The scale range is: 0 to 6 - normal/symptom absent; 7 to 19 - mild depression; 20 to 34 - moderate depression; 35 - 60 - severe depression. Reduction is a better and increase is a worse outcome.
Response rate using Montgomery-Asberg Depression Rating Scale (MADRS) at week 6. | From baseline until week 6.
  Reduction of 50% or more of the Montgomery-Asberg Depression Rating Scale (MADRS) in each patient in both interventional groups. The scale range is: 0 to 6 - normal/symptom absent; 7 to 19 - mild depression; 20 to 34 - moderate depression; 35 - 60 - severe depression. Reduction is a better and increase is a worse outcome.
Remission rate using Montgomery-Asberg Depression Rating Scale (MADRS) at week 3 | From baseline until week 3.
  Montgomery-Asberg Depression Rating Scale (MADRS) < 11 points in each patient in both interventional groups. The scale range is: 0 to 6 - normal/symptom absent; 7 to 19 - mild depression; 20 to 34 - moderate depression; 35 - 60 - severe depression. Reduction is a better and increase is a worse outcome.
Remission rate using Montgomery-Asberg Depression Rating Scale (MADRS) at week 6. | From baseline until week 6.
  Montgomery-Asberg Depression Rating Scale (MADRS) < 11 points in each patient in both interventional groups. The scale range is: 0 to 6 - normal/symptom absent; 7 to 19 - mild depression; 20 to 34 - moderate depression; 35 - 60 - severe depression. Reduction is a better and increase is a worse outcome.
Change in Hamilton Anxiety Scale (HAM-A scale) at week 3. | From baseline until week 3.
  Change in Hamilton Anxiety Scale (HAM-A scale) in each patient in both interventional groups. The outcome will be assessed by a continuous change using a mixed models statistic. The scale range is: 0-17 - mild anxiety; 18-24 moderate anxiety; 25-30 - severe anxiety. Reduction is a better and increase is a worse outcome.
Change in Hamilton Anxiety Scale (HAM-A scale) at week 6. | From baseline until week 6.
  Change in Hamilton Anxiety Scale (HAM-A scale) in each patient in both interventional groups. The outcome will be assessed by a continuous change using a mixed models statistic. The scale range is: 0-17 - mild anxiety; 18-24 moderate anxiety; 25-30 - severe anxiety. Reduction is a better and increase is a worse outcome.
Change in Global Clinical Impression Scale of Severity (GCI-S) at week 3. | From baseline until week 3.
  Change in Global Clinical Impression Scale of Severity (GCI-S) in each patient in both interventional groups. The outcome will be assessed by a continuous change using a mixed models statistic. The scale range is: 1- not sick; 2- very mild disease; 3- mild disease; 4- moderate disease; 5- intense disease; 6- severe disease; 7- extremely severe disease. Reduction is a better and increase is a worse outcome.
Change in Global Clinical Impression Scale of Severity (GCI-S) at week 6. | From baseline until week 6.
  Change in Global Clinical Impression Scale of Severity (GCI-S) in each patient in both interventional groups. The outcome will be assessed by a continuous change using a mixed models statistic. The scale range is: 1- not sick; 2- very mild disease; 3- mild disease; 4- moderate disease; 5- intense disease; 6- severe disease; 7- extremely severe disease. Reduction is a better and increase is a worse outcome.
Change in the brief version of the World Health Organization Quality of Life Questionnaire (WHOQOL-brief scale) at week 3. | From baseline until week 3.
  Change in the brief version of the World Health Organization Quality of Life Questionnaire (WHOQOL-brief scale) in both interventional groups.The scale range is: 26 to 130 points. Increase is a better and reduction is a worse outcome.
Change in the brief version of the World Health Organization Quality of Life Questionnaire (WHOQOL-brief scale) at week 6. | From baseline until week 6.
  Change in the brief version of the World Health Organization Quality of Life Questionnaire (WHOQOL-brief scale) in both interventional groups.The scale range is: 26 to 130 points. Increase is a better and reduction is a worse outcome.
Change in Global Assessment of Functioning (GAF) Scale at week 3. | From baseline until week 3.
  Change in Global Assessment of Functioning (GAF) Scale in both interventional groups. The scale range is: 1 to 100 points. Increase is a better and reduction is a worse outcome.
Change in Global Assessment of Functioning (GAF) Scale at week 6. | From baseline until week 6.
  Change in Global Assessment of Functioning (GAF) Scale in both interventional groups. The scale range is: 1 to 100 points. Increase is a better and reduction is a worse outcome.
Change in Biological Rhythm Interview of Assessment in Neuropsychiatry (BRIAN) at week 3. | From baseline until week 3.
  Change in Biological Rhythm Interview of Assessment in Neuropsychiatry (BRIAN) in both interventional groups. The scale range is: 18 to 72 points. Reduction is a better and increase is a worse outcome.
Change in Biological Rhythm Interview of Assessment in Neuropsychiatry (BRIAN) at week 6. | From baseline until week 6.
  Change in Biological Rhythm Interview of Assessment in Neuropsychiatry (BRIAN) in both interventional groups. The scale range is: 18 to 72 points. Reduction is a better and increase is a worse outcome.
Change in Barratt Impulsivity Scale of 11 items (BIS-11) at week 3. | From baseline until week 3.
  Change in Barratt Impulsivity Scale of 11 items (BIS-11) in both interventional groups. The scale range is: 30 to 120 points. Reduction is a better and increase is a worse outcome.
Change in Barratt Impulsivity Scale of 11 items (BIS-11) at week 6. | From baseline until week 6.
  Change in Barratt Impulsivity Scale of 11 items (BIS-11) in both interventional groups. The scale range is: 30 to 120 points. Reduction is a better and increase is a worse outcome.
Frequency of adverse events in UKU-SERS Scale at week 6. | From baseline until week 6.
  Frequency of adverse events in UKU-SERS Scale in both interventional groups.The scale range is: 0 to 57 points. Reduction is a better and increase is a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Moreno, PHD, Principal Investigator — University of Sao Paulo
Locations (1):
- Institute of Psychiatry, University of Sao Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Tavares DF, Suen P, Rodrigues Dos Santos CG, Moreno DH, Lane Valiengo LDC, Klein I, Borrione L, Marques Forte P, Brunoni AR, Alberto Moreno R. Treatment of mixed depression with theta-burst stimulation (TBS): results from a double-blind, randomized, sham-controlled clinical trial. Neuropsychopharmacology. 2021 Dec;46(13):2257-2265. doi: 10.1038/s41386-021-01080-9. Epub 2021 Jun 30. PMID 34193961
- [Derived] Tavares DF, Dos Santos CGR, Valiengo LDCL, Klein I, Borrione L, Forte PM, Brunoni AR, Moreno RA. Efficacy, Safety, and Tolerability of Theta-Burst Stimulation in Mixed Depression: Design, Rationale, and Objectives of a Randomized, Double-Blinded, Sham-Controlled Trial. Front Psychiatry. 2020 May 15;11:435. doi: 10.3389/fpsyt.2020.00435. eCollection 2020. PMID 32499730